CLINICAL TRIAL: NCT00836173
Title: A Phase II Study Evaluating Three Cyslces of Ifosfamide, Carboplatin, Etoposide, and Rituximab (RICE) Followed by Two Cycles of Gallium Nitrate, Rituximab and Dexamethasone (GARD) for Relapsed or Refractory Diffuse Large B-Cell Lymphoma MA
Brief Title: Rituximab, Ifosfamide, Carboplatin, and Etoposide (RICE) Followed by Gallium Nitrate, Rituximab and Dexamethasone (GARD) for Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Gallium is no longer available for the conduct of this study.
Sponsor: Loyola University (Other)
Collaborators: Genta Incorporated (Industry)
Responsible Party: Principal Investigator, Scott E Smith, MD, PhD, Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200119
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: CARBOPLATIN; DEXAMETHASONE; DIFFUSE LARGE B-CELL LYMPHOMA; ETOPOSIDE; GALLIUM NITRATE; IFOSFAMIDE; PHASE II; RELAPSED OR REFRACTORY; RITUXIMAB
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RICE followed by GARD (Experimental): 1. RICE treatment: Rituximab by intravenous infusion over 6-8 hours on day 1, Eptoposide by intravenous infusion over 2 hours on day 3-5, a 1-hour infusion of Carboplatin on day 4 and a 24-hour infusion of Ifosfamide on day 4, for 3 cycles.
  2. GaRD treatment: After RICE treatment, gallium nitrate will be given continuously over a 7 day period. In addition rituximab will be given on day 1 of each cycle. Dexamethasone will be given for the first 4 days of each cycle. The length of each cycle is 21 days.
  Interventions: Drug: RICE; Drug: GaRD Treatment

INTERVENTIONS:
Drug: RICE — RICE treatment: Rituximab by intravenous infusion over 6-8 hours on day 1, Eptoposide by intravenous infusion over 2 hours on day 3-5, a 1-hour infusion of Carboplatin on day 4 and a 24-hour infusion of Ifosfamide on day 4, each cycle is 14 days (2 weeks). Patients will receive 3 cycles of RICE treatment.
Drug: GaRD Treatment — After RICE treatment, patients will have gallium nitrate IV through a vein continuously over a 7 day period. Patients will also receive rituximab by intravenous infusion over a 3-6 hour period on day 1 of each cycle. Dexamethasone will be given as pills to be taken for 4 days in a row on the first 4 days of each cycle. The length of each cycle is 21 days (3 weeks). All patients will have 2 cycles of GaRD.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad; rituximab, ifosfamide, carboplatin and etoposide (RICE) followed by gallium nitrate, rituximab and dexamethasone (GARD) have on diffuse large B cell lymphoma.

This research is being done to try to find a more effective treatment for this type of cancer. We want to know whether treatment with rituximab, ifosfamide, carboplatin and etoposide (RICE) then followed by gallium nitrate, rituximab and dexamethasone (GARD) will improve survival.

Rituximab, ifosfamide, carboplatin and etoposide (RICE) are part of the usual treatment for diffuse large B-cell lymphoma.

Gallium nitrate, rituximab and dexamethasone (GARD) in lymphoma is experimental.

DETAILED DESCRIPTION:
This is a Phase 2 trial evaluating the efficacy of adding the combination of GaRD x 2 cycles following 3 cycles of the standard salvage regimen of RICE for the treatment of relapsed or refractory diffuse, large B-cell lymphoma (DLBCL). The study will include patients who have relapsed after 1 prior treatment regimen or who are refractory to initial chemotherapy. We will evaluate patients for response rate (both partial and complete), toxicities, as well as overall and progression free survival. Eligible patients will receive standard RICE x 3 cycles followed by GaRD x 2 cycles. Patients who would otherwise be eligible, may then proceed to autologous stem cell transplant (ASCT).

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed diffuse, large B-cell lymphoma (WHO classification diffuse large B-cell lymphoma or mediastinal large B-cell lymphoma), immunoblastic B cell lymphoma or Burkitts lymphoma. Transformed, large B-cell lymphoma will be excluded.
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with spiral CT scan.
* Must be refractory to initial therapy or have disease relapse from prior therapy and must be at least 3 weeks post treatment from prior chemotherapy or radiation therapy.
* Age >18 years.
* Life expectancy >24 weeks
* SWOG performance status <1 (Karnofsky >80%).
* Must have normal organ function (or impaired marrow function) as defined below:

  * leukocytes > or equal to 1,500/mcL
  * absolute neutrophil count >or equal to 1,000/mcL
  * platelets >or equal to 50,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT)<or equal to 2.5 X institutional upper limit of normal unless due to lymphoma involvement
  * creatinine clearance > than or equal to 60 mL/min
* Must agree not to become pregnant for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Follicular B-cell lymphomas, small lymphocytic lymphomas, chronic lymphocytic leukemia, lymphoblastic lymphomas and all T-cell lymphomas.
* Patients may not be receiving any other investigational agents, within trials in the previous 4 weeks.
* Patients with known CNS metastases are excluded from this clinical trial.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gallium nitrate, rituximab, dexamethasone, ifosfamide, carboplatin, and/or etoposide.
* Prior therapy with gallium nitrate, ifosfamide, carboplatin and/or etoposide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and women who are nursing are excluded from this study.
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with RICE and/or GaRD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine CR rates of standard salvage chemotherapy with rituximab, ifosfamide, carboplatin and etoposide (RICE) for relapsed/refractory diffuse aggressive NHL followed by a novel regimen of gallium nitrate, rituximab, and dexamethasone (GARD) | 12 weeks

SECONDARY OUTCOMES:
To determine progression-free survival and overall survival following an autologous stem cell transplant performed after the completion of the above regimen, as well as assessment of stem cell collection. | 18 months
To determine the toxicities of the regimen | approximately 12 weeks
To investigate in vitro assays that may predict response to gallium based salvage chemotherapy | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Smith, MD, PhD, FACP, Principal Investigator — Loyola University
Locations (1):
- Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois, United States